CLINICAL TRIAL: NCT00867750
Title: Radioembolisation (RE) With SIR-Spheres® Microspheres Versus Transarterial Chemoembolisation (TACE) in Patients With Unresectable Hepatocellular Carcinoma (HCC). A Comparative, Prospective, Randomised, Open, Pilot Study.
Brief Title: SIR-Spheres® Microspheres Versus Transarterial Chemoembolisation in Patients With Unresectable Hepatocellular Carcinoma
Acronym: SIRTACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SX-PHCC-001; STX0306
Record Dates: First submitted 2009-03-13; First posted 2009-03-24 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; RE; Yttrium-90; SIR-Spheres microspheres; TACE; Radioembolisation; Transarterial Chemoembolisation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RE (Experimental): Device: Radioembolisation with yttrium-90 labelled SIR-Spheres microspheres
  Interventions: Device: Radioembolisation (SIR-Spheres® microspheres)
- TACE (Active Comparator): Transarterial Chemoembolisation with embolising agent Embospheres and chemotherapeutic agent epirubicin
  Interventions: Drug: Transarterial Chemoembolisation

INTERVENTIONS:
Device: Radioembolisation (SIR-Spheres® microspheres) — Yttrium-90 SIR-Spheres microspheres
  Arms: RE
Drug: Transarterial Chemoembolisation — TACE with embolising agent Embospheres (150-300 μm or 300-500 μm diameter) with 50 mg of chemotherapeutic agent epirubicin admixed with 5 ml lipiodol.
  Arms: TACE

SUMMARY:
This study is open to patients with primary HCC who cannot be treated by potentially curative treatment modalities, such as surgical resection, liver transplantation or percutaneous ablation.

Patients that satisfy the study eligibility criteria will be randomised in a 1: 1 ratio to receive either Radioembolisation with SIR-Spheres Microspheres or the standardised Transarterial Chemoembolisation procedure.

Study Objectives

This study will evaluate and compare quality of life as well as safety and efficacy of RE or TACE in patients with unresectable HCC. Patients will be followed for a minimum of 12 months or until death wherever possible in the evaluation of the primary and secondary objectives of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged ≥ 18 years
* Unequivocal diagnosis of primary HCC (confirmed by biopsy/histology or EASL criteria)
* Tumour characteristics as follows:

  * Not more than 5 lesions
  * If single, maximal diameter ≤ 10 cm
  * If multiple, sum of maximal diameters ≤ 15 cm
  * Lesions satellite to primary tumour of less than 1 cm in maximal diameter are not included
  * At least one quantifiable lesion on hepatic MRI
* Preserved liver function, corresponding to Child-Pugh class ≤ B-7
* ECOG performance status ≤ 2
* Life expectancy ≥ 12 weeks
* Female patients of childbearing potential must have a negative pregnancy test prior to inclusion in the trial and male and female patients must agree to use an effective contraceptive method for the duration of the trial.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients expected to undergo surgery (resection or transplantation) within the 24-week period after randomisation.
* Ascites, which is detectable on physical examination or clinically symptomatic (but patients having ascites discovered by imaging only should not be excluded).
* Serum transaminases > 5 x ULN
* Lung shunt > 20%
* Extrahepatic disease
* Moderate to severe portal hypertension, as evidenced by any of the following criteria (occurring in spite of using common criteria for prophylactic treatment and therapy):

  * History of variceal haemorrhage in past 2 years
  * History of hepatic encephalopathy
  * Platelets < 50.000 /ml
  * WBC < 3.000 / ml
  * Previous TIPSS procedure
* Portal vein occlusion or hepatofugal flow.
* Impaired liver function

  * Total serum bilirubin > 2.0 mg / dL
  * Serum albumin < 3.0 g /dl
  * creatinine > 2 mg / dL
* Chemotherapy or other experimental therapy within preceding 4 weeks
* Previous TAE / TACE
* Previous radiation therapy to liver or lungs
* Contraindications for angiography (severe peripheral vascular disease or uncorrectable bleeding diathesis)
* Anatomical variants apparent on 99mTc-MAA scan precluding safe administration of RE
* Any decompensated concomitant disease
* Female patients who are pregnant, breast-feeding, or pre-menopausal and not practising efficient contraceptive method (hormonal contraceptive, intra-uterine device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life (HRQL) | 9 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS); calculated from the date of first treatment | From the date of first treatment until disease progression
Morphological tumour response; assessed using RESIST criteria | From the date of first treatment until disease progression
Functional tumour response; assessed via tumour marker reduction | From the date of first treatment until disease progression
Survival at 6 and 12 months | 6 and 12 months from the date of first treatment
Overall survival | From the date of first treatment until death
Incidence rate of portal vein invasion | From the date of first treatment until disease progression
Incidence rate of extra-hepatic disease | From the date of first treatment until disease progression
Pharmaco-economic assessment | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bruno Sangro, MD, PhD, Principal Investigator — Clinica Universitaria de Navarra; Dr. Frank Kolligs, PD, Principal Investigator — Universitäts-Klinikum München-Grosshadern
Locations (2):
- Universitäts-Klinikum München-Grosshadern, Medizinische Klinik und Poliklinik II, München, Germany
- Clinica Universitaria de Navarra, Pamplona, Spain